CLINICAL TRIAL: NCT02426476
Title: HRV Biofeedback in Pain Patients: Pilot Intervention for Pain, Fatigue & Sleep
Brief Title: HRV Biofeedback in Pain Patients
Acronym: HRVB-PP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: CLNA-006-14F
Record Dates: First submitted 2015-04-09; First posted 2015-04-27 (Estimated); Results first posted 2021-06-02 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Chronic Neuromuscular Pain
Keywords: heart rate variability; biofeedback; chronic pain; Veterans
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- active HRVB training (Experimental): Heart rate variability biofeedback training
  Interventions: Behavioral: active heart rate variability biofeedback training
- sham HRVB training (Sham Comparator): passive relaxation
  Interventions: Behavioral: sham HRVB training

INTERVENTIONS:
Behavioral: active heart rate variability biofeedback training — resonant frequency breathing, attention focusing, positive emotional state
  Other Names: a-HRVB
  Arms: active HRVB training
Behavioral: sham HRVB training — passive relaxation
  Other Names: s-HRVB
  Arms: sham HRVB training

SUMMARY:
Pain initiates a stress response that increases sympathetic output and leads to autonomic imbalance. Heart rate variability (HRV) is a easy to perform, valid measure of autonomic function. HRV biofeedback (HRV-B) is a novel biobehavioral procedure in which patients learn to restore autonomic balance by developing 'HRV Coherence'. Patients in HRV Coherence have improved mood and cognition. The investigators' pilot study showed that HRV-B alleviated chronic pain and stress among Veteran Pain Clinic patients. HRV-B thus has a pivotal role in managing pain. The proposed project is a randomized, sham-controlled, biobehavioral intervention with HRV-B to test the hypotheses that HRV-B increases HRV coherence and reduces pain, stress, fatigue, insomnia and depression and improves sleep, activity, and cognition in Veterans with chronic neuromuscular pain. The investigators hypothesize that HRV-B will (1) reduce self-reported pain and stress ratings, (2) improve objective measures of actigraphic sleep parameters (sleep latency, duration, efficiency, fragmentation), rest/activity rhythms (dichotomy index, interdaily stability) and cognitive function (reaction time, attention); and (3) alleviate self-reported fatigue and depression symptoms. Patients from two groups will be randomized to the investigators' previously established HRV-B or sham protocol (n=40 each), and will complete a baseline assessment, 6 weekly training sessions, a post-training assessment, and 4-week and 8-week follow-up evaluations post-training. Portable, hand-held, data-logging devices will be used to practice attaining HRV coherence at home by the active HRV-B training group, while those in the sham training group will get a 'stress squeeze ball'. Standard methods will quantify HRV coherence and other HRV measures, and validated instruments will be used to assess pain, stress, fatigue, insomnia, depression, and cognitive function. Wrist actigraphy will be used to objectively characterize insomnia via continuous recordings collected 24-hrs/day over three 1-week periods (pre-training, post-training, and at the 4 week follow-up assessments. Tests measuring attention and reaction time will assess changes in cognitive performance. Data analyses will apply linear models for repeated measures to evaluate the effect of HRV-B on study outcomes, and on treatment persistence, after adjusting for confounding factors. This study will be the first to examine HRV-B for pain management among Veteran chronic pain patients.

DETAILED DESCRIPTION:
This study fulfills the national Veterans Health Administration/Department of Defense (VHA/DoD) Task Force recommendation that complementary, integrative therapies for pain management be provided to Veterans. Chronic pain elicits stress which increases sympathetic output fostering autonomic nervous system imbalance, an overextended stress response, fatigue, depression and insomnia. Heart Rate Variability (HRV) is a measure of the interplay between the sympathetic and parasympathetic nervous systems, and thus is a useful and easily-measured index of autonomic balance that has a relationship to chronic pain effects. HRV biofeedback (HRV-B) is a novel, biobehavioral procedure that restores normal autonomic balance. Through HRV-B, patients increase parasympathetic cardiac output and restore autonomic balance via induction of 'HRV coherence'. The investigators' pilot study indicated that HRV-B produced coherence and alleviated self-reported ratings of chronic pain and stress among Veterans attending the investigators' Pain Clinic. The proposed clinical intervention will further test hypotheses that HRV-B increases HRV coherence, reduces self-reported pain, stress, depression, fatigue, and insomnia, and improves cognition among Veterans with chronic pain.

The specific aims are to: (1) conduct a randomized, sham-controlled, pilot intervention trial to determine whether HRV-B increases HRV coherence among chronic pain patients (n=40 each for the HRV-B and sham treatment groups; total N=80 patients); (2) determine whether HRV-B reduces self-reported pain and stress among chronic pain patients. The primary endpoints include HRV coherence, pain (Brief Pain Inventory or BPI),and stress (Perceived Stress Scale or PSS)

Outcomes will be measured at 4 time points. pre-training; post-training, one week after the 6 weekly treatments are over; at 4 weeks follow-up after post-training, and at an 8-week post-training follow-up (total time of participation is 16 weeks from pre-training to 8 week follow-up).

Furthermore, chronic stress is associated with disrupted circadian rest/activity rhythms and domains of quality of life (QoL) including fatigue, insomnia, and reduced physical and social functioning. Interventions that relieve pain thus represent a novel therapeutic target for normalizing dysfunctional rest/activity rhythms and these QoL domains among pain patients. The investigators are also interested in assessing the effects of HRV-B on cognitive function in pain patients. Thus, the investigators' secondary exploratory objectives are to determine if HRV-B: (1) improves sleep and rest/activity rhythms; (2) alleviates self-reported fatigue and depression; and (3) improves cognitive function (reaction time, attention). Circadian endpoints will be measured as actigraphic parameters of sleep (e.g., duration, efficiency), and rest/activity (e.g., dichotomy index, interdaily stability), and with the Insomnia Symptom Questionnaire (ISQ); fatigue will be assessed using the Multi-Dimensional Fatigue Inventory (MFI), which assesses general physical and mental fatigue and motivation. Depression will be assessed via the Beck Depression Inventory II (BDI-II). Cognitive function will be measured with a cognitive battery comprised of the Paced Auditory Serial Addition Test (PASAT), the Rey Auditory Verbal Learning Test (RAVLT), and the Psychomotor Vigilance Test (PVT).

Proposed Intervention. HRV-B training will follow a previously established, standardized protocol. The primary (HRV coherence, pain, stress) and exploratory outcomes (insomnia, fatigue, depression, cognition). Outcomes will be assessed at 4 time points: pre-training; post-training, one week after the 6 weekly treatments are over; at 4 weeks follow-up after post-training, and at an 8-week post-training follow-up (total time of participation is 16 weeks from pre-training to 8 week follow-up). There will be no HRV-B training at the 8 week follow-up, only assessment. Standardized procedures will characterize HRV coherence and other frequency- or time-domain HRV measures, and validated instruments will be used to assess pain and stress. Wrist actigraphy will characterize insomnia via continuous, 24-hour/day personal monitoring of rest/activity rhythms at 1-week intervals coinciding with the baseline pre-training (baseline), post-training, and 8-week follow-up assessments. The investigators will provide portable data-logging devices for practicing HRV-B at home. Sham intervention subjects will have pulse and respiration monitored but not receive active training; instead they will view a static, relaxing nature picture on a computer screen.

The investigators will control false discovery rates at 5%. Analyses will be based on intent to treat with two-sided tests. The effect of HRV-B on coherence and other HRV variables will be analyzed using linear mixed models for repeated measures data from sequential time assessments, and a between-subjects factor to evaluate the intervention after adjusting for potential confounding factors (e.g., age, standard therapy, medications, co-morbid disease). Baseline relationships between HRV and endpoints will be examined using multiple regression models. Few studies have examined the multivariate relationship between pain, autonomic dysfunction, stress, depression, sleep, rest/activity rhythms, fatigue, and cognition.

ELIGIBILITY:
Inclusion Criteria:

* are a Veteran between age 18 or older
* have chronic, non-malignant, neuro-musculoskeletal pain

Exclusion Criteria:

* a history of arrhythmia requiring medication or hospitalization
* a pacemaker or automatic implantable cardioverter-defibrillator
* a history of ischemic heart disease, heart transplant, cardiovascular surgery within 1 year
* congestive heart failure
* uncontrolled hypertension
* an active prescription for certain heart medications
* a history of seizures or use of antiseizure or anticonvulsant medication
* moderate or severe head injury or stroke
* evidence of active substance abuse or dependence (alcohol or tobacco use is not be an exclusion, participants will be asked to provide information about these behaviors in the investigators' questionnaire)
* a history of bipolar, psychotic, panic or obsessive-compulsive disorder (note: depression is an exclusion)
* cognitive impairment (dementia), neurocognitive deficits, or a central nervous system or neurological disorder (e.g., Gulf War Syndrome)
* a current or pending worker compensation claim or personal injury litigation related to the participants' symptoms

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2015-06-10 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James B Burch, Principal Investigator — Wm. Jennings Bryan Dorn VA Medical Center, Columbia, SC
Locations (1):
- Wm. Jennings Bryan Dorn VA Medical Center, Columbia, SC, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 3 patients provided informed consent and were randomized but did not show up for their baseline appointment
Period: Overall Study
Arm/Group | Active HRVB Training | Sham HRVB Training
Started | 57 | 56
Completed | 38 | 39
Not Completed | 19 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active HRVB Training | Sham HRVB Training | Total
Number analyzed (Participants) | 57 | 56 | 113
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (10) | 55 (12) | 54 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 37
  Male | 38 | 38 | 76
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 34 | 26 | 60
  White | 15 | 27 | 42
  More than one race | 8 | 3 | 11
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 57 | 56 | 113

OUTCOME MEASURES:

1. Primary Outcome: Pain Interference Rating, Measured With the Brief Pain Inventory (BPI)
Description: The BPI was developed by the World Health Organization (WHO) specifically for use among cancer patients, and it has since been widely adopted for assessment of clinical pain and pain treatment effectiveness in a variety of clinical and research settings. The possible range is 0 to 10; higher scores represent more pain interference.
Time Frame: Baseline, Week 15 (Follow-up Assessment)
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Active HRVB Training | Sham HRVB Training
Number analyzed (Participants) | 38 | 39
score on a scale
  Baseline | 7.2 [6.3 to 8.1] | 7.4 [6.3 to 8.4]
  Follow-up (week 15) | 6.2 [5.2 to 7.2] | 6.9 [5.8 to 7.9]
Statistical Analysis 1: Comparison: Active HRVB Training vs Sham HRVB Training; Linear mixed models for repeated measures (PROC MIXED in SAS) were used to assess the effects of intervention group, time, and the group by time interaction. A directional (one-sided) hypothesis was tested for the Group-by-Time interaction. The covariance matrix that minimized the Akaike Information Criterion was used. Each outcome was evaluated separately. Models were adjusted for baseline depression score and race; Test type: Superiority; p < 0.01, Mixed Models Analysis — Group by Time interaction

2. Primary Outcome: Perceived Stress Scale (PSS)
Description: The perceived stress scale measures the degree to which situations in one's life are appraised as stressful. Higher values correspond to more stress. Items were designed to assess how unpredictable, uncontrollable, and overloaded respondents find their lives. The possible range is 0-40; higher values represent more stress.
Time Frame: Baseline, Week 15 (Follow-up Assessment)
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Groups:
- HRV Biofeedback: active intervention
- Sham HRVB Training: passive relaxation control group
Arm/Group | HRV Biofeedback | Sham HRVB Training
Number analyzed (Participants) | 38 | 39
units on a scale
  Baseline | 22 [20 to 24] | 23 [21 to 25]
  Follow-up (week 15) | 20 [18 to 22] | 21 [19 to 24]
Statistical Analysis 1: Comparison: HRV Biofeedback vs Sham HRVB Training; Test type: Superiority; p = 0.87, Mixed Models Analysis — Group by Time interaction

3. Primary Outcome: Heart Rate Variability Coherence Ratio
Description: Heart rate variability coherence will allow for direct, quantitative assessment of participant performance and receipt of intervention. The HRV Coherence Ratio is obtained by identifying the maximum peak in the 0.04-0.26 Hz range of the fast Fourier transformation of heart rate interbeat intervals, then calculating the integral in a window 0.030 Hz wide centered on the highest peak in that region ('peak power', usually ~0.1 Hz), then calculating the total power of the entire spectrum. The HRV Coherence Ratio is then quantified as: peak power / (total power - peak power).
Time Frame: Baseline, Week 15 (Follow-up Assessment)
Measure: Least Squares Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Active HRVB Training | Sham HRVB Training
Number analyzed (Participants) | 38 | 39
Ratio
  Baseline | 0.18 [0.13 to 0.25] | 0.17 [0.12 to 0.25]
  Follow-up (week 15) | 0.52 [0.36 to 0.76] | 0.20 [0.13 to 0.30]
Statistical Analysis 1: Comparison: Active HRVB Training vs Sham HRVB Training; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.01, Mixed Models Analysis — Group by Time Interaction

ADVERSE EVENTS:
Time Frame: The project duration was ~4.5 years. Audits were performed annually.
Arm/Group | Active HRVB Training | Sham HRVB Training
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/57 | 1/56
Other Adverse Events (participants affected / at risk) | 1/57 | 2/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active HRVB Training (N=57) | Sham HRVB Training (N=56)
HIPAA Authorization form (Social circumstances) | 0 (0) | 1 (1) — Participant provided name or signature in only 5 of 7 locations on HIPAA Authorization form. The situation was rectified and their data was included in the analysis.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active HRVB Training (N=57) | Sham HRVB Training (N=56)
Consent form not signed by research staff (Social circumstances) | 1 (1) | 2 (2) — Research staff did not sign consent form. Participant signed both consent & HIPAA form in all 3 cases. The forms were corrected. The IRB defined these events as serious. Its uncertain whether subjects perceived this as serious.

LIMITATIONS AND CAVEATS:
The study was a behavioral intervention and is therefore not amenable to blinding.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-15): https://cdn.clinicaltrials.gov/large-docs/76/NCT02426476/Prot_SAP_000.pdf